CLINICAL TRIAL: NCT05691751
Title: Blood Loss Assessment in the Limited Application of Tourniquet During Primary Unilateral TKA: a Randomized Controlled Study
Brief Title: Blood Loss Assessment in the Limited Application of Tourniquet During Primary Unilateral TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UDMS-Orthopedics-1-2023
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Arthritis Knee; Blood Loss; Arthroplasty Complications
Keywords: total knee arthroplasty; blood loss; tourniquet; complications
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants were randomly assigned following simple randomization procedures (computerized random numbers) to 1 of 2 treatment groups, and the allocation was put into concealed envelopes independent of the surgeon and the author, and the randomization was performed by a research fellow who was not involved in patient care, the patients were blinded to the intervention during the whole period of the study, while the surgeon and the author were unblinded by opening the envelope by a research member just before initiating anesthesia, the data was collected by the author's assistant who was blinded of the intervention during the whole period of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- limited application (Experimental): Will go primary unilateral TKA with the tourniquet inflated only during cementation and final components of the prosthesis application
  Interventions: Procedure: primary unilateral total knee arthroplasty with limited application of tourniquet
- full-time application (Experimental): will go unilateral primary TKA with inflating the tourniquet prior to incision and releasing it after closure and compression bandage application
  Interventions: Procedure: primary unilateral total knee arthroplasty with full application of tourniquet

INTERVENTIONS:
Procedure: primary unilateral total knee arthroplasty with limited application of tourniquet — the tourniquet will be applicated around the proximal thigh in all patients before the incision, all patients will undergo primary unilateral TKA by the same surgeon using the medial para-patellar approach, and the prostheses used in all patients will be cruciate scarifying cemented DePuy Synthes PFC Sigma without resurfacing of the patella, intramedullary guides will be used for the femoral and tibial cuts as seen appropriate by the surgeon, however, the application time of the tourniquet during surgery will be as the allocation of each patient imply.
  Arms: limited application
Procedure: primary unilateral total knee arthroplasty with full application of tourniquet — the tourniquet will be applicated around the proximal thigh in all patients before the incision, all patients will undergo primary unilateral TKA by the same surgeon using the medial para-patellar approach, and the prostheses used in all patients will be
  Arms: full-time application

SUMMARY:
Tourniquet application in total knee arthroplasty has many benefits and might have a role in the incidence of peri-operative complications the aim of this research: is to look into the effectiveness of the limited application of tourniquet during primary unilateral total knee arthroplasty and compare the perioperative complications with the standard full-time application.

DETAILED DESCRIPTION:
Tourniquet application has been a routine choice for most joint surgeons around the world, reducing intra-operative blood loss and the better clearance of the surgical field and the better cementation technique with a blood-free cancellous bone are the main benefits, while the possible negatives are the pain of the thigh, skin burns, neurovascular complications and possibly increased risk of VTE, and the literature states a new orientation towards reducing the time of application of tourniquet or even eliminating it, favoring avoiding its risks rather than captivating its benefits so the investigator conducted a prospective randomized double-blinded controlled study, and enrolled 62 patients between the beginning of 2021 and august,2022.

after obtaining informed consent and approval by the institutional review board, the study was done in Damascus Syria, the investigator followed up every patient for six months, Participants were randomly assigned following simple randomization procedures (computerized random numbers) to 1 of 2 treatment groups, and the allocation was put into concealed envelopes independent of the surgeon and the author and the randomization was performed by a research fellow who was not involved in patient care, the tourniquet was applicated around the proximal thigh in all patients, the first group went unilateral primary TKA with inflating the tourniquet prior to incision and releasing it after closure and compression bandage application, while the second group went primary unilateral TKA with the tourniquet inflated only during cementation and final components application, the procedures were done under general, spinal or regional anesthesia based on the anesthetist consultant, a based-on-weight tranexamic acid dose was given intravenously before incision, all procedures was done by the same surgeon using the medial para-patellar approach , and the protheses used in all patients were cruciate scarifying cemented DePuy Synthes PFC Sigma without resurfacing of the patella, intramedullary guides were uses for the femoral and tibial cuts, the patients were blinded to the intervention during the whole period of the study, while the surgeon and the author were unblinded by opening the envelope by a research member just before initiating anesthesia

ELIGIBILITY:
Inclusion Criteria:

* patients between 50 and 85 years of age with end-stage knee arthritis going primary unilateral TKA after the failure of conservative treatment.

Exclusion Criteria:

* o Patients younger than 50y and older than 85y.

  * BMI less than 20 and more than 35.
  * Patients having a vascular or hematologic disease.
  * Patients who were taking anti-coagulant medicine and can't stop it.
  * Patients having acute or chronic renal failure.
  * Patients classified as the AAA as grade four or five.
  * Post-traumatic and secondary knee arthritis patients.
  * Revisions and complex primary cases.
  * Patients with an active infection or a history of lower limp infection.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
total estimated blood loss | measured once 2 days after surgery
  the total amount of lost blood in the perioperative period and will be calculated using the Gross formula which is estimated by hitting the patients' blood volume by the difference between pre and post-operative hematocrit value divided by the initial hematocrit value
intra-operative blood loss | measured once by the time of closure of the incision
  the amount of lost blood intraoperatively and will be measured by calculating the increased weight of the utilized wet mops and the volume of the suction bottle after erasing the amount of the used lavage
post-operative blood loss | measured once 2 days after surgery
  the amount of lost blood postoperatively will be calculated as the output of the drain bottle
hidden blood loss | measured once 2 days after surgery
  the amount of lost blood in the tissues that were not measured intraoperatively or postoperatively and will be calculated using the difference between total blood loss and intra and post-operative blood loss

SECONDARY OUTCOMES:
duration of surgery | measured once at the time of bandage application after closure
  the time of duration of surgery from incision to bandage application measured by minutes
surgical field clearance | measured once by the time of closure of incision
  surgical field clearance as evaluated by the surgeon
perioperative complications | assessed within two weeks intervals until 6 months after surgery
  like the incidence of infection, VTE, etc

CONTACTS AND LOCATIONS:
Overall Officials: jaber ibrahim, MD PHD, Study Chair — Damascus university - faculty of medicine - department of surgery; hakam alasaad, MD, Study Director — Damascus university - faculty of medicine - department of surgery; doried Diri, MD, Principal Investigator — Damascus university - faculty of medicine - department of surgery
Locations (1):
- Damascus university, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adie S, Harris I, Chuan A, Lewis P, Naylor JM. Selecting and optimising patients for total knee arthroplasty. Med J Aust. 2019 Feb;210(3):135-141. doi: 10.5694/mja2.12109. Epub 2019 Jan 18. PMID 30656689
- [Background] Singh JA. Epidemiology of knee and hip arthroplasty: a systematic review. Open Orthop J. 2011 Mar 16;5:80-5. doi: 10.2174/1874325001105010080. PMID 21584277
- [Background] Whittaker JL, Truong LK, Dhiman K, Beck C. Osteoarthritis year in review 2020: rehabilitation and outcomes. Osteoarthritis Cartilage. 2021 Feb;29(2):190-207. doi: 10.1016/j.joca.2020.10.005. Epub 2020 Nov 24. PMID 33242604
- [Background] Xu H, Yang J, Xie J, Huang Z, Huang Q, Cao G, Pei F. Tourniquet use in routine primary total knee arthroplasty is associated with a higher transfusion rate and longer postoperative length of stay: a real-world study. BMC Musculoskelet Disord. 2020 Sep 18;21(1):620. doi: 10.1186/s12891-020-03623-5. PMID 32948173
- [Background] Horlocker TT, Hebl JR, Gali B, Jankowski CJ, Burkle CM, Berry DJ, Zepeda FA, Stevens SR, Schroeder DR. Anesthetic, patient, and surgical risk factors for neurologic complications after prolonged total tourniquet time during total knee arthroplasty. Anesth Analg. 2006 Mar;102(3):950-5. doi: 10.1213/01.ane.0000194875.05587.7e. PMID 16492857
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Background] Vaishya R, Chauhan M, Vaish A. Bone cement. J Clin Orthop Trauma. 2013 Dec;4(4):157-63. doi: 10.1016/j.jcot.2013.11.005. Epub 2013 Dec 15. PMID 26403875
- [Background] Schroer WC, Berend KR, Lombardi AV, Barnes CL, Bolognesi MP, Berend ME, Ritter MA, Nunley RM. Why are total knees failing today? Etiology of total knee revision in 2010 and 2011. J Arthroplasty. 2013 Sep;28(8 Suppl):116-9. doi: 10.1016/j.arth.2013.04.056. Epub 2013 Aug 15. PMID 23954423
- [Background] Park JH, Restrepo C, Norton R, Mandel S, Sharkey PF, Parvizi J. Common peroneal nerve palsy following total knee arthroplasty: prognostic factors and course of recovery. J Arthroplasty. 2013 Oct;28(9):1538-42. doi: 10.1016/j.arth.2013.02.025. Epub 2013 Apr 4. PMID 23562462
- [Background] Sundaram K, Udo-Inyang I, Mont MA, Molloy R, Higuera-Rueda C, Piuzzi NS. Vascular Injuries in Total Knee Arthroplasty: A Systematic Review and Meta-Analysis. JBJS Rev. 2020 Jan;8(1):e0051. doi: 10.2106/JBJS.RVW.19.00051. PMID 32105241
- [Background] Ejaz A, Laursen AC, Kappel A, Laursen MB, Jakobsen T, Rasmussen S, Nielsen PT. Faster recovery without the use of a tourniquet in total knee arthroplasty. Acta Orthop. 2014 Aug;85(4):422-6. doi: 10.3109/17453674.2014.931197. Epub 2014 Jun 23. PMID 24954487
- [Background] Tai TW, Lin CJ, Jou IM, Chang CW, Lai KA, Yang CY. Tourniquet use in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2011 Jul;19(7):1121-30. doi: 10.1007/s00167-010-1342-7. Epub 2010 Dec 15. PMID 21161177
- [Background] Sehat KR, Evans RL, Newman JH. Hidden blood loss following hip and knee arthroplasty. Correct management of blood loss should take hidden loss into account. J Bone Joint Surg Br. 2004 May;86(4):561-5. PMID 15174554
- [Background] Gao FQ, Li ZJ, Zhang K, Sun W, Zhang H. Four Methods for Calculating Blood-loss after Total Knee Arthroplasty. Chin Med J (Engl). 2015 Nov 5;128(21):2856-60. doi: 10.4103/0366-6999.168041. PMID 26521781
- [Background] Wang C, Zhou C, Qu H, Yan S, Pan Z. Comparison of tourniquet application only during cementation and long-duration tourniquet application in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2018 Aug 30;13(1):216. doi: 10.1186/s13018-018-0927-6. PMID 30165882
- [Background] Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of a tourniquet used in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2014 Mar 6;9(1):13. doi: 10.1186/1749-799X-9-13. PMID 24602486
- [Background] Ahmed I, Chawla A, Underwood M, Price AJ, Metcalfe A, Hutchinson CE, Warwick J, Seers K, Parsons H, Wall PDH. Time to reconsider the routine use of tourniquets in total knee arthroplasty surgery. Bone Joint J. 2021 May;103-B(5):830-839. doi: 10.1302/0301-620X.103B.BJJ-2020-1926.R1. Epub 2021 Mar 8. PMID 33683139
- [Background] Cao Z, Guo J, Li Q, Wu J, Li Y. Comparison of efficacy and safety of different tourniquet applications in total knee arthroplasty: a network meta-analysis of randomized controlled trials. Ann Med. 2021 Dec;53(1):1816-1826. doi: 10.1080/07853890.2021.1991588. PMID 34726097
- [Background] Ferraris VA, Hochstetler M, Martin JT, Mahan A, Saha SP. Blood transfusion and adverse surgical outcomes: The good and the bad. Surgery. 2015 Sep;158(3):608-17. doi: 10.1016/j.surg.2015.02.027. Epub 2015 May 29. PMID 26032824
- [Background] Everhart JS, Sojka JH, Mayerson JL, Glassman AH, Scharschmidt TJ. Perioperative Allogeneic Red Blood-Cell Transfusion Associated with Surgical Site Infection After Total Hip and Knee Arthroplasty. J Bone Joint Surg Am. 2018 Feb 21;100(4):288-294. doi: 10.2106/JBJS.17.00237. PMID 29462032
- [Background] Kim C, Park SS, Davey JR. Tranexamic acid for the prevention and management of orthopedic surgical hemorrhage: current evidence. J Blood Med. 2015 Aug 25;6:239-44. doi: 10.2147/JBM.S61915. eCollection 2015. PMID 26345147
- [Background] Lu Q, Peng H, Zhou GJ, Yin D. Perioperative Blood Management Strategies for Total Knee Arthroplasty. Orthop Surg. 2018 Feb;10(1):8-16. doi: 10.1111/os.12361. Epub 2018 Feb 9. PMID 29424017